CLINICAL TRIAL: NCT06061419
Title: The Effect of Huel Powder on Appetite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2480/28560
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-06

CONDITIONS: Hunger
Keywords: Satiety; Appetite

STUDY DESIGN:
Intervention Model Description: Randomised, open label crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huel Powder (Active Comparator): This arm of the study will receive Huel as their first study meal with cornflakes and milk as their second
  Interventions: Other: Huel Powder
- Cornflakes and Milk (Active Comparator): This arm of the study will receive cornflakes and milk as their first study meal with Huel as their second
  Interventions: Other: Huel Powder

INTERVENTIONS:
Other: Huel Powder — Huel Powder v3.0 white, vanilla flavour

SUMMARY:
This project will assess the effect of Huel powdered food on the satiety of 40 generally healthy volunteers compared to a standard breakfast of cornflakes and milk.

To achieve this, we will recruit 40 (non-smoking) generally healthy volunteers to attend the study centre on two separate occasions. On each occasion they will arrive at the study centre fasted and will be given their breakfast of either Huel or Cornflakes and milk, matched for calorie content.

The aim is to identify the size and duration of any effect on satiety of the two meals.

DETAILED DESCRIPTION:
This project will assess the effect of Huel Food replacement on the satiety of 40 generally healthy volunteers compared to a standard breakfast of cornflakes and milk.

To achieve this, we will recruit 40 (non-smoking) generally healthy volunteers to attend the study centre on two separate occasions. On each occasion they will arrive at the study centre fasted and will be given their breakfast of either Huel or Cornflakes and milk, matched for calorie content.

We will ask volunteers to come to the research facility in Newcastle University, before they have had any breakfast, on two separate occasions. The volunteers must not eat or drink anything (except water) after 8 pm the evening before they come in. This includes not drinking any alcohol, tea, or coffee.

BMI, weight, and body composition (measured via electrical impedance) will also be taken at the initial visit to ensure they meet the inclusion criteria

All volunteers will be asked to complete screening questionnaires focusing on morning eating and exercise routine and the 'three factor eating' questionnaire before or during their screening visit.

A subset of volunteers (eight in total) will be recruited to collected blood samples throughout the two study visits. These volunteers will go through the same screening process but will also have their veins assessed for cannulation suitability.

During the two study visits, both sets of volunteers will be asked to complete appetite questionnaires every 15 minutes for the first hour and every 30 minutes for the remaining 3 hours.

Volunteers who have consented to provide blood samples will be asked to give samples just before they complete the appetite questionnaires.

The blood samples will be assessed for Ghrelin, CCK, PYY, Glucose, and Insulin.

All researchers are trained in GCP, phlebotomy and cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Generally Healthy
* Non-pregnant/lactating
* No known food allergies
* BMI between 20-30

Exclusion Criteria:

* Diagnosed eating disorder
* receiving regular medication (except contraceptives or statins)
* long-term illness such as high blood pressure, heart disease
* taking medication that can affect kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-29 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Hunger Visual Analogue Score | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  How hungry do you feel?
Satisfied Visual Analogue Score | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  How satisfied do you feel?
Fullness Visual Analogue Score | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  How full do you feel?
How much can you eat Visual Analogue Score | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  How much do you think you can eat?

SECONDARY OUTCOMES:
Sweet Visual Analogue Score | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Would you like to eat something sweet?
Salty Visual Analogue Score | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Would you like to eat something salty?
Savoury Visual Analogue Score | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Would you like to eat something savoury?
Fatty Visual Analogue Score | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Would you like to eat something fatty?
PYY | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Concentration of Peptide YY in plasma (pg/ml)
Ghrelin | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Concentration of Ghrelin in plasma (pg/ml)
CCK | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Concentration of Cholecystokinin in plasma (pg/ml)
Glucose | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Concentration of glucose in plasma (mmol/l)
Insulin | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes
  Concentration of Insulin in plasma (pmol/l)

IPD SHARING:
Plan to Share IPD: No